CLINICAL TRIAL: NCT07299760
Title: Evaluation of the Analgesic Efficacy of Parasternal Block and Parasternal Plus Serratus Anterior Plane Block in Patients Undergoing Coronary Artery Bypass Grafting Surgery
Brief Title: Analgesic Efficacy of Parasternal Block Versus Parasternal Plus Serratus Anterior Plane Block After Coronary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ekin Guran, MD, Attending anesthesiologist, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PS_SAPB
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Bypass Grafting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Parasternal Block (Active Comparator): After induction of general anaesthesia and before skin incision, an ultrasound-guided bilateral parasternal intercostal plane block will be performed.
  Interventions: Procedure: parasternal block
- Arm B: Serratus Anterior Plane Block (Experimental): In addition to the bilateral parasternal block described for the comparator arm, patients randomized to the experimental arm will receive an ultrasound-guided bilateral serratus anterior plane block.
  Interventions: Procedure: parasternal block; Procedure: parasternal block + serratus anterior plane block

INTERVENTIONS:
Procedure: parasternal block — After induction of general anaesthesia and before skin incision, an ultrasound-guided bilateral parasternal intercostal plane block will be performed. A linear ultrasound probe will be placed parasagittally at the 2nd and 4th intercostal spaces approximately 2-3 cm lateral to the sternum. A block needle will be advanced in-plane beneath the pectoralis major muscle and above the internal intercostal muscles, and local anaesthetic (0.25% bupivacaine) will be injected bilaterally. Total dose will not exceed 2 mg/kg. Postoperative systemic analgesia (patient-controlled analgesia) will be identical in both groups.
Procedure: parasternal block + serratus anterior plane block — In addition to the bilateral parasternal block described for the comparator arm, patients randomized to the experimental arm will receive an ultrasound-guided bilateral serratus anterior plane block. With the patient in supine position, the linear ultrasound probe will be placed over the 6th rib in the anterior axillary line. The needle will be advanced in-plane beneath the serratus anterior muscle and above the rib, and 0.25% bupivacaine will be injected into the fascial plane on each side. The combined total dose of local anaesthetic for both blocks will not exceed 2 mg/kg. Postoperative systemic analgesia will be identical in both groups.
  Arms: Arm B: Serratus Anterior Plane Block

SUMMARY:
This single-centre randomized clinical trial will compare two regional anaesthesia techniques for postoperative pain control in adult patients undergoing elective coronary artery bypass grafting (CABG) with sternotomy. All patients will receive a bilateral parasternal block as part of routine multimodal analgesia. Patients will be randomized to receive either parasternal block alone or a combination of parasternal block and serratus anterior plane block. The primary objective is to evaluate whether adding a serratus anterior plane block improves postoperative pain scores compared with parasternal block alone. Secondary objectives include comparing opioid consumption, need for rescue analgesics, opioid-related side effects, and length of stay in the intensive care unit and hospital.

DETAILED DESCRIPTION:
Background: Postoperative pain after coronary artery bypass surgery arises from both the sternotomy incision and the chest tube insertion sites and may impair mobilisation, deep breathing, and coughing. Fascial plane blocks of the chest wall, such as parasternal block and serratus anterior plane block, are increasingly used because they are technically simple and have a low complication risk. Previous observational data suggested that combining bilateral parasternal block and serratus anterior plane block provides effective analgesia after CABG, but sample size was small and no randomized comparison has been performed.

Objectives: The primary objective is to compare postoperative pain intensity between parasternal block alone and parasternal plus serratus anterior plane block in adult patients undergoing elective CABG with sternotomy. Secondary objectives are to compare total opioid consumption (tramadol via patient-controlled analgesia), need for rescue analgesics, incidence of opioid-related adverse events (e.g. nausea and vomiting), and intensive care unit and hospital length of stay between the two groups.

Methods: This is a prospective, randomized, parallel-group, low-risk interventional study conducted in the Anaesthesiology and Reanimation Department of Ankara Etlik City Hospital. Adult patients (≥18 years) scheduled for elective coronary bypass surgery due to coronary artery disease and classified as ASA II-IV will be screened for eligibility. After induction of general anaesthesia and before surgical incision, all patients will receive an ultrasound-guided bilateral parasternal block. Patients randomized to the experimental arm will additionally receive a bilateral serratus anterior plane block. Local anaesthetic dosing will follow routine clinical practice, with a total dose not exceeding 2 mg/kg of 0.25% bupivacaine. All patients will receive 40 ml of 0.25% bupivacaine. The parasternal group will receive a bilateral parasternal block via administering 20 ml of 0.25% bupivacaine bilaterally. The parasternal+serratus anterior plane block group will receive 10 ml of 0.25% bupivacaine to bilateral parasternal and deep serratus planes.

Pain intensity will be assessed using the Numeric Rating Scale (NRS, 0-10) at extubation (T0) and postoperative 4, 6, 12, and 24 hours (T4, T6, T12, T24). Postoperative analgesia will include standard intravenous acetaminophen and tramadol via patient-controlled analgesia; total tramadol dose (demand and delivered), rescue analgesic requirement, and adverse events will be recorded in the first 24 postoperative hours.

Sample size: Based on a two-group comparison with an effect size of 0.6, α = 0.0,5, and β = 0.2, 72 patients are required to achieve 80% power.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* American Society of Anesthesiologists (ASA) physical status III-IV
* Scheduled for elective coronary artery bypass grafting surgery with sternotomy for coronary artery disease
* Able to provide written informed consent

Exclusion Criteria

* Allergy or contraindication to local anaesthetic agents
* Minimally invasive bypass surgery or off-pump procedures planned
* Emergency cardiac surgery
* Preoperative Numeric Rating Scale (NRS) pain score ≥ 3
* Chronic opioid use in the preoperative period
* Infection or structural abnormality at planned block sites
* Any condition preventing postoperative pain assessment or PCA use (e.g. severe cognitive impairment)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Total Tramadol Consumption | 24-hour post-extubation
  Cumulative dose of tramadol (mg) delivered by patient-controlled analgesia (PCA) in the first 24 hours post-extubation

SECONDARY OUTCOMES:
Resting Numeric Rating Scale (NRS) Pain Score | 24 hour post-extubation
  NRS score during rest (0= no pain, 10= worst imaginable pain)
Dynamic Numeric Rating Scale (NRS) Pain Score | 24-hour post-extubation
  NRS score during coughing or deep inspiration (0= no pain, 10= worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik City Hospital, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the primary publication may be shared upon reasonable request to the principal investigator after publication of the results.
Supporting Information: Study Protocol, ICF
Time Frame: De-identified individual participant data underlying the primary publication may be shared upon reasonable request to the principal investigator after publication of the results.
Access Criteria: De-identified individual participant data underlying the primary publication may be shared upon reasonable request to the principal investigator after publication of the results.

REFERENCES:
- [Result] Zengin EN, Yigit H, Cobas M, Salman N, Asli Demir Z. The analgesic effects of combined bilateral parasternal block and serratus anterior plane block for coronary artery bypass grafting surgery. BMC Anesthesiol. 2024 Aug 5;24(1):274. doi: 10.1186/s12871-024-02659-7. PMID 39103782